CLINICAL TRIAL: NCT02291679
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Parallel-group Trial of Linaclotide (72 ug or 145 ug) Administered Orally for 12 Weeks to Patients With Chronic Idiopathic Constipation
Brief Title: Trial of Linaclotide in Patients With Chronic Idiopathic Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ironwood Pharmaceuticals, Inc. (Industry)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MCP-103-309
Record Dates: First submitted 2014-11-11; First posted 2014-11-14 (Estimated); Results first posted 2017-05-19 (Actual); Last update posted 2017-06-15 (Actual); Status verified 2017-05

CONDITIONS: Chronic Idiopathic Constipation
MeSH Terms: interventions — linaclotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 72 μg linaclotide (Experimental): 72 μg oral linaclotide, once daily for 12 weeks
  Interventions: Drug: Linaclotide
- 145 μg linaclotide (Experimental): 145 μg oral linaclotide, once daily for 12 weeks
  Interventions: Drug: Linaclotide
- Placebo (Placebo Comparator): matching placebo, once daily for 12 weeks
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: Linaclotide
  Other Names: Linzess; Constella
  Arms: 145 μg linaclotide; 72 μg linaclotide
Drug: Matching Placebo
  Arms: Placebo

SUMMARY:
The objective of this trial was to determine the efficacy and safety of linaclotide 72 ug administered once daily to patients with chronic idiopathic constipation (CIC). The primary efficacy parameter is the percentage of participants in each dosing group that meet the protocol definition for complete spontaneous bowel movement (CSBM) Overall Responder.

DETAILED DESCRIPTION:
The trial also included a 145 ug linaclotide treatment arm (an FDA-approved dose for CIC) as an established positive control to validate the study design.

ELIGIBILITY:
Inclusion Criteria:

* Patient has completed a colonoscopy if one is needed according to the American Gastroenterological Association (AGA) criteria, with no clinically significant findings
* Patient has no clinically significant findings on a physical examination and clinical laboratory tests
* Patient meets protocol criteria for CIC: reports < 3 bowel movements (BMs) per week and reports one or more of the following during ≥ 25% of BMs: straining, lumpy or hard stools, sensation of incomplete evacuation during the 3 months before the diagnosis with the onset at least 6 months before the diagnosis
* Patient is compliant with daily interactive voice response system (IVRS) calls
* Patient reports an average of < 3 complete spontaneous BMs (CSBMs) and ≤ 6 SBMs per week by the IVRS over the 14 calendar days before the Randomization Visit and the calendar day of Randomization.

Exclusion Criteria:

* Patient has history of loose or watery stools
* Patient has symptoms of or been diagnosed with irritable bowel syndrome (IBS)
* Patient has a structural abnormality of the gastrointestinal (GI) tract or a disease or condition that can affect GI motility
* Patient has any protocol-excluded or clinically significant medical or surgical history that could confound the study assessments
* Patient has Bristol Stool Form Scale score of 7 during Pretreatment period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1223 (Actual)
Dates: Start 2014-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard J Lavins, MD, Study Chair — Ironwood Pharmaceuticals, Inc.
Locations (84):
- United States (84):
  - Ironwood Investigational Site, Huntsville, Alabama
  - Ironwood Investigational Site, Phoenix, Arizona
  - Ironwood Investigational Site, Tucson, Arizona
  - Ironwood Investigational Site, North Little Rock, Arkansas
  - Ironwood Investigational Site, Anaheim, California
  - Ironwood Investigational Site, Chula Vista, California
  - Ironwood Investigational Site, Garden Grove, California
  - Ironwood Investigational Site, La Mesa, California
  - Ironwood Investigational Site, North Hollywood, California
  - Ironwood Investigational Site, Orange, California
  - Ironwood Investigational Site, San Diego, California
  - Ironwood Investigational Site, Thousand Oaks, California
  - Ironwood Investigational Site, Colorado Springs, Colorado
  - Ironwood Investigational Site, Bristol, Connecticut
  - Ironwood Investigational Site, Boynton Beach, Florida
  - Ironwood Investigational Site, Coral Gables, Florida
  - Ironwood Investigational Site, DeLand, Florida
  - Ironwood Investigational Site, Hialeah, Florida
  - Ironwood Investigational Site, Inverness, Florida
  - Ironwood Investigational Site, Jupiter, Florida
  - Ironwood Investigational Site, Kissimmee, Florida
  - Ironwood Investigational Site, Lauderdale Lakes, Florida
  - Ironwood Investigational Site, Miami, Florida
  - Ironwood Investigational Site, Orlando, Florida
  - Ironwood Investigational Site, Ormond Beach, Florida
  - Ironwood Investigational Site, Port Orange County, Florida
  - Ironwood Investigational Site, South Miami, Florida
  - Ironwood Investigational Site, Tampa, Florida
  - Ironwood Investigational Site, West Palm Beach, Florida
  - Ironwood Investigational Site, Winter Park, Florida
  - Ironwood Investigational Site, Atlanta, Georgia
  - Ironwood Investigational Site, Oakwood, Georgia
  - Ironwood Investigational Site, Sandy Springs, Georgia
  - Ironwood Investigational Site, Evansville, Indiana
  - Ironwood Investigational Site, Bastrop, Louisiana
  - Ironwood Investigational Site, Metairie, Louisiana
  - Ironwood Investigational Site, Shreveport, Louisiana
  - Ironwood Investigational Site, Baltimore, Maryland
  - Ironwood Investigational Site, Chevy Chase, Maryland
  - Ironwood Investigational Site, Hagerstown, Maryland
  - Ironwood Investigational Site, Hollywood, Maryland
  - Ironwood Investigational Site, Boston, Massachusetts
  - Ironwood Investigational Site, Wellesley, Massachusetts
  - Ironwood Investigational Site, Chesterfield, Michigan
  - Ironwood Investigational Site, Troy, Michigan
  - Ironwood Investigational Site, Wyoming, Michigan
  - Ironwood Investigational Site, Jackson, Mississippi
  - Ironwood Investigational Site, St Louis, Missouri
  - Ironwood Investigational Site, Bozeman, Montana
  - Ironwood Investigational Site, Las Vegas, Nevada
  - Ironwood Investigational Site, Brooklyn, New York
  - Ironwood Investigational Site, Endwell, New York
  - Ironwood Investigational Site, Great Neck, New York
  - Ironwood Investigational Site, Charlotte, North Carolina
  - Ironwood Investigational Site, Greensboro, North Carolina
  - Ironwood Investigational Site, High Point, North Carolina
  - Ironwood Investigational Site, Lenoir, North Carolina
  - Ironwood Investigational Site, Raleigh, North Carolina
  - Ironwood Investigational Site, Wilmington, North Carolina
  - Ironwood Investigational Site, Winston-Salem, North Carolina
  - Ironwood Investigational Site, Fargo, North Dakota
  - Ironwood Investigational Site, Cincinnati, Ohio
  - Ironwood Investigational Site, Columbus, Ohio
  - Ironwood Investigational Site, Mentor, Ohio
  - Ironwood Investigational Site, Sylvania, Ohio
  - Ironwood Investigational Site, Oklahoma City, Oklahoma
  - Ironwood Investigational Site, Levittown, Pennsylvania
  - Ironwood Investigational Site, Anderson, South Carolina
  - Ironwood Investigational Site, Greer, South Carolina
  - Ironwood Investigational Site, Simpsonville, South Carolina
  - Ironwood Investigational Site, Dakota Dunes, South Dakota
  - Ironwood Investigational Site, Bristol, Tennessee
  - Ironwood Investigational Site, Chattanooga, Tennessee
  - Ironwood Investigational Site, Knoxville, Tennessee
  - Ironwood Investigational Site, Beaumont, Texas
  - Ironwood Investigational Site, Dallas, Texas
  - Ironwood Investigational Site, El Paso, Texas
  - Ironwood Investigational Site, Houston, Texas
  - Ironwood Investigational Site, Longview, Texas
  - Ironwood Investigational Site, San Antonio, Texas
  - Ironwood Investigational Site, South Ogden, Utah
  - Ironwood Investigational Site, Christiansburg, Virginia
  - Ironwood Investigational Site, Lynchburg, Virginia
  - Ironwood Investigational Site, La Crosse, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 2244 participants were screened; 1223 were randomized and 1021 were not randomized (478 participants were screen failures and 543 participants were pretreatment failures).
Period: Overall Study
Arm/Group | Placebo | 72 μg Linaclotide | 145 μg Linaclotide
Started | 401 | 411 | 411
Completed | 357 | 369 | 352
Not Completed | 44 | 42 | 59
Not completed — Adverse Event | 2 | 12 | 19
Not completed — Protocol Violation | 5 | 1 | 7
Not completed — Withdrew Consent | 18 | 10 | 15
Not completed — Lost to Follow-up | 12 | 10 | 9
Not completed — Insufficient Therapeutic Response | 5 | 5 | 7
Not completed — Other | 2 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 72 μg Linaclotide | 145 μg Linaclotide | Total
Number analyzed (Participants) | 401 | 411 | 411 | 1223
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (14.7) | 45.8 (14.3) | 46.8 (14.0) | 46.0 (14.3)
Age, Customized [Count of Participants; unit: Participants]
  18 to < 40 years | 142 | 140 | 128 | 410
  40 to < 65 years | 220 | 235 | 240 | 695
  ≥ 65 years | 39 | 36 | 43 | 118
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 316 | 312 | 314 | 942
  Male | 85 | 99 | 97 | 281
Complete Spontaneous Bowel Movement Weekly Rate [Mean (Standard Deviation); unit: CSBMs/week] — Number of complete spontaneous bowel movements (CSBMs) per week. A CSBM is defined as a spontaneous bowel movement (SBM) that is associated with a sense of complete evacuation. An SBM is defined as a bowel movement (BM) that occurred in the absence of laxative, enema, or suppository use on either the calendar day of the BM or the calendar day before the BM. Baseline efficacy values are derived from the interactive voice response system (IVRS) daily diary data collected in the Pretreatment Period, specifically the period of time from 14 days before randomization up to the time of randomization.
  CSBMs/week | 0.25 (0.48) | 0.22 (0.52) | 0.20 (0.44) | 0.22 (0.48)
Spontaneous Bowel Movement Weekly Rate [Mean (Standard Deviation); unit: SBMs/week] — Number of spontaneous bowel movements (SBMs) per week. An SBM is defined as a BM that occurred in the absence of laxative, enema, or suppository use on either the calendar day of the BM or the calendar day before the BM. Baseline efficacy values are derived from the IVRS daily diary data collected in the Pretreatment Period, specifically the period of time from 14 days before randomization up to the time of randomization.
  SBMs/week | 1.56 (1.15) | 1.74 (1.42) | 1.67 (1.38) | 1.66 (1.33)
Stool Consistency Score [Mean (Standard Deviation); unit: units on a scale] — Measured daily using the 7-point ordinal Bristol Stool Form Scale (BSFS; 1=separate hard lumps like nuts [difficult to pass]; 2=sausage shaped but lumpy; 3=like a sausage but with cracks on surface; 4=like a sausage or snake, smooth and soft; 5=soft blobs with clear-cut edges [passed easily]; 6=fluffy pieces with ragged edges, a mushy stool; 7=watery, no solid pieces [entirely liquid]). Baseline efficacy values are derived from the IVRS daily diary data collected in the Pretreatment Period, specifically the period of time from 14 days before randomization up to the time of randomization. Population: Participants who did not have an SBM at baseline had missing Stool Consistency baseline scores.
  units on a scale
    number analyzed (Participants) | 359 | 360 | 364 | 1083
    (all) | 2.04 (1.02) | 1.94 (0.93) | 1.96 (0.94) | 1.98 (0.96)
Straining Score [Mean (Standard Deviation); unit: units on a scale] — Straining was measured daily using a 5-point ordinal scale (1 = not at all; 2 = a little bit; 3 = a moderate amount; 4 = a great deal; 5 = an extreme amount). Baseline efficacy values are derived from the IVRS daily diary data collected in the Pretreatment Period, specifically the period of time from 14 days before randomization up to the time of randomization. Population: Participants who did not have an SBM at baseline had missing Straining baseline scores.
  units on a scale
    number analyzed (Participants) | 359 | 360 | 364 | 1083
    (all) | 3.51 (0.88) | 3.62 (0.86) | 3.52 (0.82) | 3.55 (0.85)
Abdominal Discomfort [Mean (Standard Deviation); unit: units on a scale] — Abdominal discomfort was measured daily using an 11-point numerical rating scale (NRS; 0 = none; 10 = very severe). Baseline efficacy values are derived from the IVRS daily diary data collected in the Pretreatment Period, specifically the period of time from 14 days before randomization up to the time of randomization.
  units on a scale | 4.76 (2.56) | 4.64 (2.74) | 4.71 (2.66) | 4.70 (2.65)
Abdominal Bloating [Mean (Standard Deviation); unit: units on a scale] — Abdominal bloating was measured daily using an 11-point NRS (0 = none; 10 = very severe). Baseline efficacy values are derived from the IVRS daily diary data collected in the Pretreatment Period, specifically the period of time from 14 days before randomization up to the time of randomization.
  units on a scale | 5.29 (2.39) | 5.24 (2.61) | 5.30 (2.57) | 5.27 (2.52)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of 12-Week CSBM Overall Responders
Description: A 12-week CSBM Overall Responder is a participant who was a CSBM Weekly Responder for at least 9 of the 12 weeks of the Treatment Period. A CSBM Weekly Responder is a participant who had a CSBM weekly frequency rate that was 3 or greater and increased by 1 or more from baseline, and completed ≥ 4 IVRS calls for the specified week.
  A CSBM is defined as an SBM that is associated with a sense of complete evacuation. An SBM is defined as a bowel movement BM that occurred in the absence of laxative, enema, or suppository use on either the calendar day of the BM or the calendar day before the BM.
Time Frame: Week 12
Population: Intent-to-Treat Population: all randomized participants who received at least one dose of study drug. Only data for the 72 μg dose versus placebo arms were prospectively defined and evaluated as a primary endpoint; per protocol, data for the 145 μg dose arm were not collected for any pre-specified primary or secondary outcome measures.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 72 μg Linaclotide
Number analyzed (Participants) | 401 | 411
percentage of participants
  Responder | 4.7 | 13.4
  Non-Responder | 95.3 | 86.6
Statistical Analysis 1: Comparison: Placebo vs 72 μg Linaclotide; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value is obtained from the Cochran-Mantel-Haenszel (CMH) tests controlling for baseline SBM stratum and geographic region; Odds Ratio (OR) = 3.03, 95% CI 2-sided [1.76 to 5.20] — Placebo as reference. Odds ratio and 95% confidence interval (CI) for the odds ratio are obtained from the CMH tests controlling for baseline SBM stratum and geographic region

2. Secondary Outcome: Change From Baseline in 12-Week CSBM Frequency Rate
Description: A participant's 12-week CSBM Frequency Rate is the CSBM rate (CSBMs/week) calculated over the 12 weeks of the Treatment Period. A CSBM is defined as an SBM that is associated with a sense of complete evacuation. An SBM is defined as a BM that occurred in the absence of laxative, enema, or suppository use on either the calendar day of the BM or the calendar day before the BM.
Time Frame: Baseline, Week 1 to Week 12
Population: Intent-to-Treat Population: all randomized participants who received at least one dose of study drug. Only data for the 72 μg dose versus placebo arms were prospectively defined and evaluated as a secondary endpoint; data for the 145 μg dose arm were defined and evaluated as an additional endpoint per protocol.
Measure: Least Squares Mean (Standard Error); unit: CSBMs/week
Arm/Group | Placebo | 72 μg Linaclotide
Number analyzed (Participants) | 401 | 411
CSBMs/week | 0.884 (0.142) | 1.725 (0.139)
Statistical Analysis 1: Comparison: Placebo vs 72 μg Linaclotide; Test type: Superiority; p < 0.0001, ANCOVA — P-value is based on a pairwise comparison versus placebo in an ANCOVA model with treatment group, baseline SBM stratum, and geographic region as factors and baseline value as covariate; LS Mean Difference = 0.841, 95% CI 2-sided [0.505 to 1.176] — Linaclotide - Placebo. Estimate and 95% CI are based on a least squares (LS) mean difference from an ANCOVA model with treatment group, baseline SBM stratum, and geographic region as factors and baseline value as covariate

3. Secondary Outcome: Change From Baseline in 12-Week SBM Frequency Rate
Description: A participant's 12-week SBM Frequency Rate is the SBM rate (SBMs/week) calculated over the 12-weeks of the Treatment Period. An SBM is defined as a BM that occurred in the absence of laxative, enema, or suppository use on either the calendar day of the BM or the calendar day before the BM.
Time Frame: Baseline, Week 1 to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: SBMs/week
Arm/Group | Placebo | 72 μg Linaclotide
Number analyzed (Participants) | 401 | 411
SBMs/week | 1.329 (0.169) | 2.366 (0.166)
Statistical Analysis 1: Comparison: Placebo vs 72 μg Linaclotide; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 1.037, 95% CI 2-sided [0.636 to 1.438] — Linaclotide - Placebo. Estimate and 95% CI are based on a LS mean difference from an ANCOVA model with treatment group, baseline SBM stratum, and geographic region as factors and baseline value as covariate

4. Secondary Outcome: Change From Baseline in 12-Week Stool Consistency Score
Description: Stool consistency was measured daily using the 7-point ordinal Bristol Stool Form Scale (BSFS; 1 = separate hard lumps like nuts [difficult to pass]; 2 = sausage shaped but lumpy; 3 = like a sausage but with cracks on surface; 4 = like a sausage or snake, smooth and soft; 5 = soft blobs with clear-cut edges [passed easily]; 6 = fluffy pieces with ragged edges, a mushy stool; 7 = watery, no solid pieces [entirely liquid]). The participant's BSFS score for the Treatment Period is the average of the non-missing BSFS scores from the SBMs reported by the participant during the 12-week Treatment Period.
Time Frame: Baseline, Week 1 to Week 12
Population: Intent-to-Treat Population: all randomized participants who received ≥ 1 dose of study drug and reported an SBM during the Baseline period. Only data for the 72 μg dose versus placebo arms were prospectively defined and evaluated as a secondary endpoint; data for the 145 μg dose arm were defined and evaluated as an additional endpoint per protocol.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 72 μg Linaclotide
Number analyzed (Participants) | 344 | 349
units on a scale | 1.065 (0.076) | 1.693 (0.074)
Statistical Analysis 1: Comparison: Placebo vs 72 μg Linaclotide; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.628, 95% CI 2-sided [0.450 to 0.806] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Change From Baseline in 12-Week Straining Score
Description: Straining was measured daily using a 5-point ordinal scale (1 = not at all; 2 = a little bit; 3 = a moderate amount; 4 = a great deal; 5 = an extreme amount). The participant's straining score for the Treatment Period is the average of the non-missing straining scores from the SBMs reported by the participant during the 12-week Treatment Period.
Time Frame: Baseline, Week 1 to Week 12
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 72 μg Linaclotide
Number analyzed (Participants) | 344 | 349
units on a scale | -0.789 (0.051) | -1.118 (0.050)
Statistical Analysis 1: Comparison: Placebo vs 72 μg Linaclotide; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.329, 95% CI 2-sided [-0.449 to -0.210] — [estimate comment as in outcome 3, analysis 1]

6. Secondary Outcome: Percentage of 12-Week CSBM Overall Responders (>1 SBM/Week Subpopulation)
Description: A 12-week CSBM Overall Responder is a participant who was a CSBM Weekly Responder for at least 9 of the 12 weeks of the Treatment Period. A CSBM Weekly Responder is a participant who had a CSBM weekly frequency rate that was 3 or greater and increased by 1 or more from baseline, and completed ≥4 IVRS calls for the specified week.
  A CSBM is defined as an SBM that is associated with a sense of complete evacuation. An SBM is defined as a BM that occurred in the absence of laxative, enema, or suppository use on either the calendar day of the BM or the calendar day before the BM.
Time Frame: Week 12
Population: Participants in the Intent-to-Treat Population who reported >1 SBM/week during the Pretreatment Period (14 days prior to randomization). Only data for the 72 μg dose versus placebo arms were prospectively defined and evaluated as a secondary endpoint; data for the 145 μg dose arm were defined and evaluated as an additional endpoint per protocol.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 72 μg Linaclotide
Number analyzed (Participants) | 226 | 244
percentage of participants
  Responder | 7.1 | 17.2
  Non-Responder | 92.9 | 82.8
Statistical Analysis 1: Comparison: Placebo vs 72 μg Linaclotide; Test type: Superiority; p = 0.0008, Cochran-Mantel-Haenszel — P-value is obtained from the CMH tests controlling for geographic region; Odds Ratio (OR) = 2.68, 95% CI 2-sided [1.47 to 4.87] — Placebo as reference. Odds ratio and 95% CI for the odds ratio are obtained from the CMH tests controlling for geographic region

7. Secondary Outcome: Percentage of Month 1 CSBM Responders
Description: A Month 1 CSBM Responder is a participant who is a CSBM weekly responder for at least 3 of the 4 weeks of Month 1 of the Treatment Period. A CSBM weekly responder is a participant who had a CSBM weekly frequency rate that was 3 or greater and increased by 1 or more from baseline based on a minimum of 4 complete IVRS calls for that week.
  A CSBM is defined as an SBM that is associated with a sense of complete evacuation. An SBM is defined as a BM that occurred in the absence of laxative, enema, or suppository use on either the calendar day of the BM or the calendar day before the BM.
Time Frame: Month 1
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 72 μg Linaclotide
Number analyzed (Participants) | 401 | 411
percentage of participants
  Responder | 6.2 | 14.8
  Non-Responder | 93.8 | 85.2
Statistical Analysis 1: Comparison: Placebo vs 72 μg Linaclotide; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value is obtained from the CMH tests controlling for geographic region and baseline stratum; Odds Ratio (OR) = 2.58, 95% CI 2-sided [1.58 to 4.20] — Placebo as reference. Odds ratio and 95% CI for the odds ratio are obtained from the CMH tests controlling for geographic region and baseline stratum

8. Secondary Outcome: Percentage of Month 2 CSBM Responders
Description: A Month 2 CSBM Responder is a participant who is a CSBM weekly responder for at least 3 of the 4 weeks of Month 2 of the Treatment Period. A CSBM weekly responder is a participant who had a CSBM weekly frequency rate that was 3 or greater and increased by 1 or more from baseline based on a minimum of 4 complete IVRS calls for that week.
  A CSBM is defined as an SBM that is associated with a sense of complete evacuation. An SBM is defined as a BM that occurred in the absence of laxative, enema, or suppository use on either the calendar day of the BM or the calendar day before the BM.
Time Frame: Month 2
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 72 μg Linaclotide
Number analyzed (Participants) | 401 | 411
percentage of participants
  Responder | 9.5 | 18.7
  Non-Responder | 90.5 | 81.3
Statistical Analysis 1: Comparison: Placebo vs 72 μg Linaclotide; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel — P-value is obtained from the CMH tests controlling for geographic region and baseline stratum; Odds Ratio (OR) = 2.15, 95% CI 2-sided [1.42 to 3.26] — [estimate comment as in outcome 7, analysis 1]

9. Secondary Outcome: Percentage of Month 3 CSBM Responders
Description: A Month 3 CSBM Responder is a participant who is a CSBM weekly responder for at least 3 of the 4 weeks of Month 3 of the Treatment Period. A CSBM weekly responder is a participant who had a CSBM weekly frequency rate that was 3 or greater and increased by 1 or more from baseline based on a minimum of 4 complete IVRS calls for that week.
  A CSBM is defined as an SBM that is associated with a sense of complete evacuation. An SBM is defined as a BM that occurred in the absence of laxative, enema, or suppository use on either the calendar day of the BM or the calendar day before the BM.
Time Frame: Month 3
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 72 μg Linaclotide
Number analyzed (Participants) | 401 | 411
percentage of participants
  Responder | 14.2 | 20.2
  Non-Responder | 85.8 | 79.8
Statistical Analysis 1: Comparison: Placebo vs 72 μg Linaclotide; Test type: Superiority; p = 0.0342, Cochran-Mantel-Haenszel — P-value is obtained from the CMH tests controlling for geographic region and baseline stratum; Odds Ratio (OR) = 1.49, 95% CI 2-sided [1.03 to 2.17] — [estimate comment as in outcome 7, analysis 1]

10. Secondary Outcome: Change From Baseline in 12-Week Abdominal Bloating
Description: Abdominal bloating was measured daily using an 11-point NRS (0 = none; 10 = very severe). The participant's abdominal bloating score for the Treatment Period is the average of the non-missing daily participant assessments of abdominal bloating scores reported during the 12-week Treatment Period.
Time Frame: Baseline, Week 1 to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 72 μg Linaclotide
Number analyzed (Participants) | 401 | 411
units on a scale | -1.052 (0.097) | -1.372 (0.095)
Statistical Analysis 1: Comparison: Placebo vs 72 μg Linaclotide; Test type: Superiority; p = 0.0063, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.319, 95% CI 2-sided [-0.548 to -0.090] — [estimate comment as in outcome 3, analysis 1]

11. Secondary Outcome: Change From Baseline in 12-Week Abdominal Discomfort
Description: Abdominal discomfort was measured daily using an 11-point NRS (0 = none; 10 = very severe). The participant's abdominal discomfort score for the Treatment Period is the average of the non-missing daily participant assessments of abdominal discomfort scores reported during the 12-week Treatment Period.
Time Frame: Baseline, Week 1 to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 72 μg Linaclotide
Number analyzed (Participants) | 401 | 411
units on a scale | -1.146 (0.090) | -1.323 (0.089)
Statistical Analysis 1: Comparison: Placebo vs 72 μg Linaclotide; Test type: Superiority; p = 0.1028, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.178, 95% CI 2-sided [-0.391 to 0.036] — [estimate comment as in outcome 3, analysis 1]

12. Other Pre Specified Outcome: Percentage of 12-Week CSBM Overall Sustained Responders
Description: A 12-week CSBM Overall Sustained Responder is a participant who was a CSBM Weekly Responder for at least 9 of the 12 weeks of the Treatment Period, including ≥ 3 of the last 4 weeks. A CSBM Weekly Responder is a participant who had a CSBM weekly frequency rate that was 3 or greater and increased by 1 or more from baseline, and completed ≥ 4 IVRS calls for the specified week.
  A CSBM is defined as an SBM that is associated with a sense of complete evacuation. An SBM is defined as a BM that occurred in the absence of laxative, enema, or suppository use on either the calendar day of the BM or the calendar day before the BM.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 72 μg Linaclotide
Number analyzed (Participants) | 401 | 411
percentage of participants
  Responder | 4.7 | 12.4
  Non-Responder | 95.3 | 87.6
Statistical Analysis 1: Comparison: Placebo vs 72 μg Linaclotide; Test type: Superiority; p = 0.0001, Cochran-Mantel-Haenszel — P-value is obtained from the CMH tests controlling for baseline SBM stratum and geographic region; Odds Ratio (OR) = 2.78, 95% CI 2-sided [1.61 to 4.80] — Placebo as reference. Odds ratio and 95% CI for the odds ratio are obtained from the CMH tests controlling for baseline SBM stratum and geographic region

ADVERSE EVENTS:
Time Frame: From first dose of double-blind study drug up to Week 12/End of Treatment Visit (Day 85 + 3 days) for nonserious events and within 30 days of the date of last dose of double-blind study drug for serious events.
Arm/Group | Placebo | 72 μg Linaclotide | 145 μg Linaclotide
Serious Adverse Events (participants affected / at risk) | 4/401 | 3/411 | 2/411
Other Adverse Events (participants affected / at risk) | 28/401 | 79/411 | 91/411
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=401) | 72 μg Linaclotide (N=411) | 145 μg Linaclotide (N=411)
Colitis (Gastrointestinal disorders) | 0 | 1 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Azotaemia (Renal and urinary disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=401) | 72 μg Linaclotide (N=411) | 145 μg Linaclotide (N=411)
Diarrhea (Gastrointestinal disorders) | 28 | 79 | 91

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI may publish or disclose the results of the study 24 months after final data lock provided that sponsor can review the publication prior to public release, sponsor can request removal of confidential information of sponsor (not including results of trial), and sponsor can request a publication delay in order to protect potentially patentable information. Furthermore, if a publication committee is developing an initial publication, PI is to delay disclosure until that publication is published.